CLINICAL TRIAL: NCT02353286
Title: Endoscopic Treatment of Benign Biliary Strictures and Cystic Duct Leakages With a Novel Biodegradable Polydioxanone Biliary Stent
Brief Title: Endoscopic Treatment of Benign Biliary Strictures and Cystic Duct Leakages With a Novel Biodegradable Biliary Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Antti Siiki, MD, Tampere University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biodegradable Biliary stent
Record Dates: First submitted 2015-01-16; First posted 2015-02-02 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Biliary Tract Diseases
Keywords: Biodegradable stents, ERCP
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post-cholecystecomy bile leak (Experimental): Endoscopic insertion of biodegradable biliary stent
  Interventions: Device: Endoscopic insertion of biodegradable biliary stent
- Benign biliary stricture (Experimental): Endoscopic insertion of biodegradable biliary stent
  Interventions: Device: Endoscopic insertion of biodegradable biliary stent

INTERVENTIONS:
Device: Endoscopic insertion of biodegradable biliary stent — Endoscopic insertion of biodegradable biliary stent
  Other Names: Braided, self-expanding polydioxanone stent, Ella, Czech Rep

SUMMARY:
Patients with either post-cholecystectomy bile leak or benign biliary stricture are recruited for endoscopic insertion of a biodegradable biliary stent. A follow-up of 12 months with repeated serum samples and magnetic resonance imaging is scheduled. The primary end points are feasibility of endoscopic insertion with the novel implantation device and stricture or leak resolution as well as clinical treatment success.

DETAILED DESCRIPTION:
Benign biliary strictures (BBS) and post-cholecystectomy bile leaks have traditionally been treated endoscopically with plastic stents. In BBS, promising results of covered self-expanding metal stent use have been recently published. However, in both BBS and post-cholecystectomy bile leak the need of stent therapy is temporary and endoscopic stent exchange or removal is unavoidable. These two groups of patients may be the ones that would most obviously benefit from biodegradable (BD) biliary stents. Studies of BD stents on animal models have shown excellent long term patency and safety both in biliary and pancreatic duct as well better outcome compared to plastic stents after post-cholecystectomy bile leak in an animal study. Until recently, non-operative insertion of BD polydioxanone stent in human biliary tract has been possible only via percutaneous route.

With the novel implantation device, the BD stents (braided, self-expanding polydioxanone stent, 8 x 40-60mm, Ella, Czech republic) may be used endoscopically during endoscopic retrograde cholangio-pancreatography (ERCP).

The hypothesis is that larger diameter and radial expansion strength provide at least similar treatment success as the current method of endoscopic insertion of plastic or covered self-expanding metal stents in bile leak and BBS, respectively. However, later stent exchange or removal is not necessary with BD stents.

ELIGIBILITY:
Inclusion Criteria:

* informed-consent patients with diagnosed or suspected post-cholecystectomy biliary leak or benign biliary stricture.

Exclusion Criteria:

* Patients with contra-indications for magnetic resonance imaging (MRI) or surgically altered gastro-duodenal anatomy (e.g. roux-y-loop) are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical treatment success of stricture or leakage, treatment failure rate measured by change in treatment protocol or unplanned interventions, radiologic stricture diameter in MRI, radiologic stent degradation in MRI | The follow-up of 12 months after stent implantation
  Stent patency, unplanned admissions and interventions, signs of cholangitis during treatment assessed by repeated liver function tests, magnetic resonance imaging and interview. Change in stent diameter and gradual radiologic dissappearance due to degradation assessed by repeated MRI and liver function tests, stricture resolution assessed by repeated MRI and radiologic measurement of stricture width as well as liver function tests, leakage resolution assessed by disappearance of biliary fluid collection in MRI and liver function tests

SECONDARY OUTCOMES:
ERCP complications, late adverse events during stent therapy | 30 days from stent implantation, late adverse events up to 12 months
  endoscopic retrograde cholangio-pancreatography (ERCP) and stent implantation related complications graded mild-moderate-severe according to Cotton et al 1991, unplanned admissions and incidence of late adverse events such as acute cholangitis until up to 12 months of follow-up assessed by repeated MRI, phone interview, blood samples and review of patient records at each follow-up contact.
Technical success of stent insertion | intraoperative
  To assess the usefulness and safety of a novel endoscopic implantation device measured by success rate of stent implantation and evaluation possible intra-procedural technical challenges during ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Laukkarinen, Md, PhD, Study Director — Dept. of Gastroenterology and Alimentary Tract Surgery; Juhani Sand, Md, PhD, Study Director — Dept. of Gastroenterology and Alimentary Tract Surgery
Locations (1):
- Tampere University Hospital, Dept. of Gastroenterology and Alimentary Tract Surgery, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mauri G, Michelozzi C, Melchiorre F, Poretti D, Tramarin M, Pedicini V, Solbiati L, Cornalba G, Sconfienza LM. Biodegradable biliary stent implantation in the treatment of benign bilioplastic-refractory biliary strictures: preliminary experience. Eur Radiol. 2013 Dec;23(12):3304-10. doi: 10.1007/s00330-013-2947-2. Epub 2013 Jul 11. PMID 23842947
- [Background] Laukkarinen J, Nordback I, Mikkonen J, Karkkainen P, Sand J. A novel biodegradable biliary stent in the endoscopic treatment of cystic-duct leakage after cholecystectomy. Gastrointest Endosc. 2007 Jun;65(7):1063-8. doi: 10.1016/j.gie.2006.11.059. PMID 17531643
- [Background] Grolich T, Crha M, Novotny L, Kala Z, Hep A, Necas A, Hlavsa J, Mitas L, Misik J. Self-expandable biodegradable biliary stents in porcine model. J Surg Res. 2015 Feb;193(2):606-12. doi: 10.1016/j.jss.2014.08.006. Epub 2014 Aug 9. PMID 25201575
- [Background] Lorenzo-Zuniga V, Moreno-de-Vega V, Marin I, Boix J. Biodegradable stents in gastrointestinal endoscopy. World J Gastroenterol. 2014 Mar 7;20(9):2212-7. doi: 10.3748/wjg.v20.i9.2212. PMID 24605020
- [Derived] Siiki A, Rinta-Kiikka I, Sand J, Laukkarinen J. A pilot study of endoscopically inserted biodegradable biliary stents in the treatment of benign biliary strictures and cystic duct leaks. Gastrointest Endosc. 2018 Apr;87(4):1132-1137. doi: 10.1016/j.gie.2017.10.042. Epub 2017 Nov 8. PMID 29128386
- [Derived] Siiki A, Rinta-Kiikka I, Sand J, Laukkarinen J. Biodegradable biliary stent in the endoscopic treatment of cystic duct leak after cholecystectomy: the first case report and review of literature. J Laparoendosc Adv Surg Tech A. 2015 May;25(5):419-22. doi: 10.1089/lap.2015.0068. Epub 2015 Apr 8. PMID 25853929